CLINICAL TRIAL: NCT01319058
Title: Laser or Debrider Tonsillotomy Versus Monopolar Tonsillectomy in Obstructive Sleep Apnea; Inflammation as a Determinate of Outcome
Brief Title: Outcome of Laser or Debrider Tonsillotomy Versus Tonsillectomy in Obstructive Sleep Apnea
Acronym: TVLOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Ben-Zion Joshua, MD, Soroka University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: sor495810ctil
Record Dates: First submitted 2011-03-17; First posted 2011-03-21 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; Tonsillectomy; Tonsillotomy; Inflammation; Pain; Post tonsillectomy bleeding
MeSH Terms: conditions — Sleep Apnea, Obstructive; Inflammation; Pain | interventions — Tonsillectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Electrocautery tonsillectomy (Active Comparator): Children undergoing tonsillectomy and adenoidectomy for obstructive sleep apnea
  Interventions: Procedure: Tonsillectomy, laser tonsillotomy, debrider tonsillotomy
- Debrider tonsillotomy (Active Comparator): Children undergoing debrider tonsillotomy + adenoidectomy for obstructive sleep apnea.
  Interventions: Procedure: Tonsillectomy, laser tonsillotomy, debrider tonsillotomy
- Laser tonsillotomy (Active Comparator): Children undergoing laser tonsillotomy + adenoidectomy for obstructive sleep apnea.
  Interventions: Procedure: Tonsillectomy, laser tonsillotomy, debrider tonsillotomy

INTERVENTIONS:
Procedure: Tonsillectomy, laser tonsillotomy, debrider tonsillotomy — Each arm will be treated by one of the three methods in addition to adenoidectomy

SUMMARY:
Tonsil surgery for children suffering from obstructive sleep apnea have significant post operative morbidity including pain and occasionally bleeding. This morbidity is partly caused by post surgical inflammation. This inflammatory process can be quantified using various proinflammatory cytokines.

the goal of this study is to objectively compare the inflammatory process after treatment of obstructive sleep apnea with different surgical approaches to the enlarged tonsils.

DETAILED DESCRIPTION:
Tonsil surgery for children suffering from obstructive sleep apnea have significant post operative morbidity including pain and occasionally bleeding. This morbidity is partly caused by post surgical inflammation. This inflammatory process can be quantified using various proinflammatory cytokines.

the goal of this study is to objectively compare the inflammatory process after treatment of obstructive sleep apnea with different surgical approaches to the enlarged tonsils.

In the study three approaches are prospectively compared:

1. Tonsillectomy - using electrocautery resecting all tonsillar tissue.
2. Debrider Tonsillotomy - reducing the tonsillar tissue with a debrider.
3. laser Tonsillotomy - reducing tonsillar tissue using a CO2 laser.

All patients will be randomized to one of three arms. Each arm will include 25 children.

All children will have a preoperative and postoperative sleep study. Questioners assessing pain, amount of medication used to control pain and sleep disturbance during the first 7 days after surgery will be filled by the child caretaker.

Blood will be drawn immediately before surgery and 18-24 hours after surgery. The following blood products will be assessed: White blood cells, clotting factors, C reactive protein, IL1 beta,TNF alpha, IL6, IL2.

If the study will show objectively and subjectively that partial resection of the tonsil compared to complete tonsillectomy is less painful and has less postoperative inflammation.

ELIGIBILITY:
Inclusion Criteria:

age 2-16 obstructive sleep apnea AHI>5 Hypertrophy of tonsils and adenoids

-

Exclusion Criteria:

Children with recurrent tonsillitis craniofacial anomalies Neuromuscular disease Down syndrome

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2010-08; Primary Completion 2013-01 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Difference between the three arms regarding serum IL1 beta, TNF alpha, IL2, IL6. | 12 months

SECONDARY OUTCOMES:
Difference between the three arms regarding pain, post tonsillectomy bleeding and post operative sleep disturbance. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Marc M Puterman, MD, Principal Investigator — Soroka University Medical Center; Aviv D Goldbart, MD, Study Director — Soroka University Medical Center
Locations (1):
- Soroka Hospital, Beersheba, Israel

REFERENCES:
- [Background] Friedman BC, Hendeles-Amitai A, Kozminsky E, Leiberman A, Friger M, Tarasiuk A, Tal A. Adenotonsillectomy improves neurocognitive function in children with obstructive sleep apnea syndrome. Sleep. 2003 Dec 15;26(8):999-1005. doi: 10.1093/sleep/26.8.999. PMID 14746381
- [Background] Ericsson E, Lundeborg I, Hultcrantz E. Child behavior and quality of life before and after tonsillotomy versus tonsillectomy. Int J Pediatr Otorhinolaryngol. 2009 Sep;73(9):1254-62. doi: 10.1016/j.ijporl.2009.05.015. Epub 2009 Jun 17. PMID 19539380
- [Background] Anand A, Vilela RJ, Guarisco JL. Intracapsular versus standard tonsillectomy: review of literature. J La State Med Soc. 2005 Sep-Oct;157(5):259-61. PMID 16374970
- [Derived] Blackshaw H, Springford LR, Zhang LY, Wang B, Venekamp RP, Schilder AG. Tonsillectomy versus tonsillotomy for obstructive sleep-disordered breathing in children. Cochrane Database Syst Rev. 2020 Apr 29;4(4):CD011365. doi: 10.1002/14651858.CD011365.pub2. PMID 32347984